CLINICAL TRIAL: NCT02943395
Title: Color Stability of E.Max CAD Laminate Veneers Cemented With Light Cure Versus Dual Cure Amine Free Adhesive Resin Cement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mahmoud hossam eldin elkomy, dentist at egyption ministry of health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17191405
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Tooth Discoloration
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- dual cure amine free adhesive resin cement (Experimental): resin cement that get activated by both light and chemicals
  Interventions: Other: E.Max CAD Laminate Veneers cemented with dual cure amine free adhesive resin cement
- light cured adhesive resin cement (Active Comparator): resin cement that only get activated by light
  Interventions: Other: E.Max CAD Laminate Veneers cemented with light cured adhesive resin cement

INTERVENTIONS:
Other: E.Max CAD Laminate Veneers cemented with dual cure amine free adhesive resin cement
  Arms: dual cure amine free adhesive resin cement
Other: E.Max CAD Laminate Veneers cemented with light cured adhesive resin cement
  Arms: light cured adhesive resin cement

SUMMARY:
Light curing cements used for laminate veneers may be not totally cured in certain areas, so dual cured resin cements may solve this problem yet the dual cured cements containing amines cause yellowish discoloration of the veneers after time.

A new dual cured cement which is amine free is introduced so the investigators have to try it clinically using parallel groups in randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to be:

* From 18-60 years old, and able to read and sign the informed consent document
* physically and psychologically able to tolerate conventional restorative procedures
* Have no active periodontal or pulpal diseases, have teeth with good restorations
* Patients with teeth problems indicated for laminate veneer (e.g. discoloration, fracture not involve more than 50% enamel loss, mild malposition, ….)
* Willing to return for follow-up examinations and evaluation

Exclusion Criteria:

* Patients in the growth stage with partially erupted teeth
* Patient with fractured teeth of more than 50% enamel loss
* Patients with poor oral hygiene and motivation
* Pregnant women
* Psychiatric problems or unrealistic expectations
* Lack of opposite occluding dentition in the area intended for restoration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Color stability assessed clinically using easy shade vita device | 1 Year
  Color stability

SECONDARY OUTCOMES:
Patient satisfaction assessed using a Questionnaire | 1 Year
  Questionnaire for the patient satisfaction

REFERENCES:
- [Background] Magalhaes AP, Cardoso Pde C, de Souza JB, Fonseca RB, Pires-de-Souza Fde C, Lopez LG. Influence of activation mode of resin cement on the shade of porcelain veneers. J Prosthodont. 2014 Jun;23(4):291-5. doi: 10.1111/jopr.12098. Epub 2013 Oct 7. PMID 24118675
- [Background] Gresnigt MM, Kalk W, Ozcan M. Clinical longevity of ceramic laminate veneers bonded to teeth with and without existing composite restorations up to 40 months. Clin Oral Investig. 2013 Apr;17(3):823-32. doi: 10.1007/s00784-012-0790-5. Epub 2012 Jul 21. PMID 22821429